CLINICAL TRIAL: NCT04425018
Title: MARGetuximab Or Trastuzumab (MARGOT): A Phase II Study Comparing Neoadjuvant Paclitaxel/Margetuximab/Pertuzumab to Paclitaxel/Trastuzumab/Pertuzumab in Patients With Stage II-III HER2-positive Breast Cancer
Brief Title: MARGetuximab Or Trastuzumab (MARGOT)
Acronym: MARGOT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: MacroGenics (Industry); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Principal Investigator, Adrienne G. Waks, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-068
Record Dates: First submitted 2020-04-15; First posted 2020-06-11 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; pertuzumab; margetuximab; Trastuzumab; Ogivri

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paclitaxel + Pertuzumab + Margetuximab (Experimental): The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits.Cycle=21 days
  * Paclitaxel- via IV, Day 1,8,15 of each cycle
  * Margetuximab via IV, Day 1 of each cycle
  * Pertuzumab via IV, Day 1 of each cycle
  Interventions: Drug: Paclitaxel; Drug: Pertuzumab; Drug: Margetuximab
- Paclitaxel + Pertuzumab + Trastuzumab (Experimental): The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits.Cycle=21 days
  * Paclitaxel- via IV, Day 1,8,15 of each cycle
  * Pertuzumab via IV, Day 1 of each cycle
  * Trastuzumab via IV, Day 1 of each cycle
  Interventions: Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Paclitaxel — Pre-determined dose administered via IV, Day 1,8,15 of each cycle 4 study cycles, or 12 weeks.
  Other Names: Taxol; Onxal
Drug: Pertuzumab — Pre-determined dose administered via IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
  Other Names: Perjeta
Drug: Margetuximab — Pre-determined dose administered by IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
  Other Names: Margenza
  Arms: Paclitaxel + Pertuzumab + Margetuximab
Drug: Trastuzumab — Pre-determined dose administered via IV Day 1 of each 21- day cycle for 4 study cycles, or 12 weeks.
  Other Names: Herceptin; Kanjinti; Ogivri; Herzuma
  Arms: Paclitaxel + Pertuzumab + Trastuzumab

SUMMARY:
The purpose of this study is to determine how well participants with stage II-III HER2-positive breast cancer respond to pre-operative treatment using one of two different combinations of drugs.

Drugs and Combinations used:

* Paclitaxel, Pertzumab and Margetuximab (Margenza)
* Paclitaxel, Pertzumab and Trastuzumab (Herceptin)

DETAILED DESCRIPTION:
This is a randomized open-label phase II trial comparing paclitaxel/margetuximab/pertuzumab (TMP) to paclitaxel/trastuzumab/pertuzumab (THP) in patients with anatomic stage II-III HER2 positive breast cancer.

* The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits.
* Participants will be randomized, which means randomly assigned, to one of two treatment arms. The treatment arms in this study and the names of the study drugs in each arm are:

  * Arm A: Paclitaxel, Pertzumab and Margetuximab
  * Arm B: Paclitaxel, Pertzumab and Trastuzumab

Participants will receive study treatment for 12 weeks prior to surgery and will be followed for 10 years after surgery. After surgery, some participants will continue to receive the study drug margetuximab for a year in total, if they respond very well to the first 12 weeks of treatment with margetuximab.

It is expected that about 171 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

The FDA (the U.S. Food and Drug Administration) has approved paclitaxel, trastuzumab (Herceptin), and pertuzumab as part of a pre-operative treatment option for stage II-III HER2-positive breast cancer.

The U.S. Food and Drug Administration (FDA) has approved margetuximab (Margenza) for advanced HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III (according to AJCC cancer staging manual anatomic staging table, 8th edition) histologically confirmed invasive carcinoma of the breast. A minimum tumor size of 1.5 cm (in breast mass or axillary lymph node) determined by physical exam or imaging (whichever is larger) is required. Patients with inflammatory breast carcinoma (T4d) are NOT eligible.
* Centrally confirmed to have a low affinity CD16 germline genotype (FF or FV)
* HER-2 positive by 2018 American Society of Clinical Oncology/College of American Pathologists criteria, as assessed by standard institutional guidelines (central testing is not required).
* ER/PR determination is required. ER- and PR-assays should be performed by immunohistochemical methods according to standard institutional guidelines
* Bilateral breast cancers are allowed as long as both cancers are HER2-positive (as defined in 3.1.2), or the contralateral cancer is a <1 cm, ER+ tumor.
* Patients with multifocal or multicentric disease are eligible if the treating investigator hasdetermined the patient should be treated as HER2-positive.
* Breast imaging should include dedicated ultrasound of the ipsilateral axilla. For subjects with a clinically positive axilla based on exam or imaging, a fine needle aspiration or core biopsy procedure will be performed to determine the presence of metastatic disease in the lymph nodes (though lymph node sampling procedure need not be resulted prior to patient's registration on trial, as long as all other eligibility are met).
* Men and women (with any menopausal status) ≥18 years of age are eligible.
* ECOG performance status 0 or 1
* Required laboratory values demonstrating adequate organ function:

  * ANC ≥ 1000/mm3
  * Hemoglobin ≥ 9 g/dl
  * Platelets ≥ 100,000/mm3
  * Serum creatinine < 1.5 x ULN (institutional) OR calculated GFR ≥ 60mL/min
  * Total bilirubin ≤ 1.5 x ULN (institutional). For patients with Gilbert Syndrome, the direct bilirubin should be within the institutional normal range OR total bilirubin ≤ 2.0 mg/dL.
  * AST and ALT ≤ 2.5x ULN (institutional) Left ventricular ejection fraction (LVEF) ≥ 50%.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of treatment start. Childbearing potential is defined as: those who have not been surgically sterilized and/or have had a menstrual period in the past 12 months
* Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 7 months after the last dose of study treatment.
* Patients with a history of ipsilateral or contralateral DCIS or LCIS are eligible.
* Patients undergoing breast conservation therapy (i.e. lumpectomy) must not have any contraindications to radiation therapy.
* Non-English-speaking patients are eligible but will be exempt from patient-completed questionnaires.
* Willing and able to sign informed consent.
* Willing to undergo breast biopsy for research purposes.

Exclusion Criteria:

* Pregnant or nursing women due to the teratogenic potential of the study drugs.
* Active, unresolved infection requiring intervention
* Receipt of intravenous antibiotics for infection within 7 days prior to registration.
* Uncontrolled hypertension (systolic >180 mm Hg and/or diastolic >100 mm Hg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication, unstable angina, congestive heart failure (CHF) of New York Heart Association (NYHA) Class II or higher, or serious cardiac arrhythmia requiring medication.
* Significant symptoms (Grade ≥ 2) from peripheral neuropathy.
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness, uncontrolled infections, uncontrolled diabetes.
* Any prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation, or experimental therapy.
* Patients with any prior history of invasive breast cancer within the past 5 years are not eligible. Non-metastatic invasive breast cancers diagnosed more than 5 years ago and any other type of prior non-metastatic cancer is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2027-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (14):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Brigham Cancer Center - Foxborough, Foxborough, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Dana-Farber at South Shore Hospital, Weymouth, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - UPMC Hillman Cancer Center - Arnold Palmer at Mountain View, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center - Arnold Palmer at Norwin, Irwin, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine Medical Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Fred Hutchinson Cancer Care, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Pertuzumab + Margetuximab: The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits.Cycle=21 days
  * Paclitaxel- via IV, Day 1,8,15 of each cycle
  * Margetuximab via IV, Day 1 of each cycle
  * Pertuzumab via IV, Day 1 of each cycle
  Paclitaxel: Pre-determined dose administered via IV, Day 1,8,15 of each cycle 4 study cycles, or 12 weeks.
  Pertuzumab: Pre-determined dose administered via IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
  Margetuximab: Pre-determined dose administered by IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
- Paclitaxel + Pertuzumab + Trastuzumab: The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits.Cycle=21 days
  * Paclitaxel- via IV, Day 1,8,15 of each cycle
  * Pertuzumab via IV, Day 1 of each cycle
  * Trastuzumab via IV, Day 1 of each cycle
  Paclitaxel: Pre-determined dose administered via IV, Day 1,8,15 of each cycle 4 study cycles, or 12 weeks.
  Pertuzumab: Pre-determined dose administered via IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
  Trastuzumab: Pre-determined dose administered via IV Day 1 of each 21- day cycle for 4 study cycles, or 12 weeks.
Period: Overall Study
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Started | 118 | 56
Completed | 117 | 54
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients who received at least one dose of their assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab | Total
Number analyzed (Participants) | 117 | 54 | 171
Age, Continuous [Median (Full Range); unit: Years] | 52.1 [30.4 to 79.7] | 55.1 [31.5 to 76.0] | 52.6 [30.4 to 79.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 54 | 171
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 6 | 22
  Not Hispanic or Latino | 99 | 46 | 145
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 90 | 42 | 132
  Race: Black or African American | 13 | 4 | 17
  Race: Asian | 5 | 2 | 7
  Race: Other | 9 | 6 | 15
Clinical stage of primary breast cancer [Count of Participants; unit: Participants]
  Stage II | 100 | 46 | 146
  Stage III | 17 | 8 | 25
Hormone receptor status of primary breast cancer [Count of Participants; unit: Participants]
  Positive (ER >= 1% or PR >= 1%) | 74 | 37 | 111
  Negative (ER < 1% and PR < 1%) | 43 | 17 | 60
CD16A Genotype [Count of Participants; unit: Participants] — The Fc-gamma RIIIA (CD16) stimulatory receptor is encoded by two alleles that differ at amino acid 158: a V allele (valine; higher affinity) and an F allele (phenylalanine; lower affinity)
  Participants
    FF | 50 | 30 | 80
    FV | 67 | 24 | 91

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: Compare the percentage of pathologic complete response (pCR) between patients treated with neoadjuvant TMP versus THP. Subject was considered a pCR responder if they achieved RCB 0 (no residual disease at surgery) and did not receive any additional non-protocol neoadjuvant treatment. Subject was considered a pCR non-responder if they did not achieve RCB 0 (RCB I, II, or III, or did not receive surgery) or if they received additional non-protocol neoadjuvant therapy.
  RCB is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to 3, defined using established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB). Higher RCB score indicates more tumor burden remaining, thus worse outcome. RCB in this trial was determined according to local pathology review.
Time Frame: 12 weeks
Population: Subjects who received at least one dose of their assigned treatment and were deemed eligible for the study based on all listed inclusion and exclusion criteria. Note: One subject in "Paclitaxel + Pertuzumab + Margetuximab" arm was excluded from pCR analysis because they were diagnosed with inflammatory breast cancer (IBC) after starting treatment, and IBC was an exclusion criteria of the study (this reduced the number of analyzed participants in this arm from 117 to 116).
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 116 | 54
Participants
  pCR Responder | 65 | 24
  pCR Non-Responder | 51 | 30
Statistical Analysis 1: Comparison: Paclitaxel + Pertuzumab + Margetuximab vs Paclitaxel + Pertuzumab + Trastuzumab; Test type: Superiority; p = 0.188, Fisher Exact; Risk Difference (RD) = 11.6, 95% CI 2-sided [-5.8 to 29.0] — Estimate and corresponding Wald 95% confidence interval of the difference in pCR response rates (%) between the "Paclitaxel + Pertuzumab + Margetuximab" and "Paclitaxel + Pertuzumab + Trastuzumab" arms

2. Secondary Outcome: Rate of Pathologic Complete Response in Hormone Receptor Positive (HR+) Subjects
Description: In hormone receptor positive (HR+) patients, compare the rate of pathologic complete response (pCR) between patients treated with neoadjuvant TMP versus THP. Subject was considered a pCR responder if they achieved RCB 0 (no residual disease at surgery) and did not receive any additional non-protocol neoadjuvant treatment. Subject was considered a pCR non-responder if they did not achieve RCB 0 (RCB I, II, or III, or did not receive surgery) or if they received additional non-protocol neoadjuvant therapy.
  RCB is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to 3, defined using established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB). Higher RCB score indicates more tumor burden remaining, thus worse outcome. RCB in this trial was determined according to local pathology review.
Time Frame: 12 weeks
Population: Hormone receptor positive (HR+) subjects with hormone receptor positive (HR+) primary breast cancers who received at least one dose of their assigned treatment and were deemed eligible for the study based on all listed inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 74 | 37
Participants
  pCR Responder | 40 | 13
  pCR Non-Responder | 34 | 24
Statistical Analysis 1: Comparison: Paclitaxel + Pertuzumab + Margetuximab vs Paclitaxel + Pertuzumab + Trastuzumab; Test type: Superiority; p = 0.0715, Fisher Exact; Risk Difference (RD) = 18.9, 95% CI 2-sided [-2.2 to 40.1] — Estimate and corresponding Wald 95% confidence interval of the difference in pCR response rates (%) between the "Paclitaxel + Pertuzumab + Margetuximab" and "Paclitaxel + Pertuzumab + Trastuzumab" arms among HR+ subjects

3. Secondary Outcome: Rate of Pathologic Complete Response in Hormone Receptor Negative (HR-) Subjects
Description: In hormone receptor negative (HR-) patients, compare the rate of pathologic complete response (pCR) between patients treated with neoadjuvant TMP versus THP. Subject was considered a pCR responder if they achieved RCB 0 (no residual disease at surgery) and did not receive any additional non-protocol neoadjuvant treatment. Subject was considered a pCR non-responder if they did not achieve RCB 0 (RCB I, II, or III, or did not receive surgery) or if they received additional non-protocol neoadjuvant therapy.
  RCB is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to 3, defined using established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB). Higher RCB score indicates more tumor burden remaining, thus worse outcome. RCB in this trial was determined according to local pathology review.
Time Frame: 12 weeks
Population: HR- subjects who received at least one dose of their assigned treatment and were deemed eligible for the study based on all listed inclusion and exclusion criteria. Note: One subject in "Paclitaxel + Pertuzumab + Margetuximab" arm was excluded from pCR analysis because they were diagnosed with inflammatory breast cancer (IBC) after starting treatment, and IBC was an exclusion criteria of the study (this reduced the number of analyzed participants in this arm from 43 to 42).
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 42 | 17
Participants
  pCR Responder | 25 | 11
  pCR Non-Responder | 17 | 6
Statistical Analysis 1: Comparison: Paclitaxel + Pertuzumab + Margetuximab vs Paclitaxel + Pertuzumab + Trastuzumab; Test type: Superiority; p = 0.7754, Fisher Exact; Risk Difference (RD) = -5.2, 95% CI 2-sided [-36.5 to 26.1] — Estimate and corresponding Wald 95% confidence interval of the difference in pCR response rates (%) between the "Paclitaxel + Pertuzumab + Margetuximab" and "Paclitaxel + Pertuzumab + Trastuzumab" arms among HR- subjects

4. Secondary Outcome: Residual Cancer Burden (RCB) Scores
Description: Assess Residual Cancer Burden (RCB) scores in patients treated with TMP or THP, reported using the Residual Cancer Burden calculator from M.D Anderson.
  RCB is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to 3, defined using established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB). Higher RCB score indicates more tumor burden remaining, thus worse outcome. RCB in this trial was determined according to local pathology review.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 116 | 54
Participants
  RCB-0 (no residual disease) | 65 | 24
  RCB-I (minimal residual disease) | 8 | 7
  RCB-II (moderate residual disease) | 29 | 15
  RCB-III (extensive residual disease) | 2 | 1
  Received additional neoadjuvant therapy | 10 | 7
  Surgery not performed | 2 | 0

5. Secondary Outcome: Residual Cancer Burden (RCB) Scores in Hormone Receptor Positive (HR+) Subjects
Description: Among hormone receptor positive (HR+) patients, assess Residual Cancer Burden (RCB) scores in patients treated with TMP or THP, reported using the Residual Cancer Burden calculator from M.D Anderson.
Time Frame: 12 weeks
Population: Hormone receptor positive (HR+) subjects who received at least one dose of their assigned treatment and were deemed eligible for the study based on all listed inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 74 | 37
Participants
  RCB-0 (no residual disease) | 40 | 13
  RCB-I (minimal residual disease) | 7 | 4
  RCB-II (moderate residual disease) | 21 | 13
  RCB-III (extensive residual disease) | 1 | 1
  Received additional neoadjuvant therapy | 5 | 6
  Surgery not performed | 0 | 0

6. Secondary Outcome: Residual Cancer Burden (RCB) Scores in Hormone Receptor Negative (HR-) Subjects
Description: Among hormone receptor negative (HR-) subjects, assess Residual Cancer Burden (RCB) scores in patients treated with TMP or THP, reported using the Residual Cancer Burden calculator from M.D Anderson.
  RCB is used to assess the response to neoadjuvant chemotherapy in breast cancer patients and is in a scale of 0 to 3, defined using established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB). Higher RCB score indicates more tumor burden remaining, thus worse outcome. RCB in this trial was determined according to local pathology review.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 42 | 17
Participants
  RCB-0 (no residual disease) | 25 | 11
  RCB-I (minimal residual disease) | 1 | 3
  RCB-II (moderate residual disease) | 8 | 2
  RCB-III (extensive residual disease) | 1 | 0
  Received additional neoadjuvant therapy | 5 | 1
  Surgery not performed | 2 | 0

7. Secondary Outcome: Dose-limiting Toxicities (DLTs) in theTMP Arm (Paclitaxel/Margetuximab/Pertuzumab) During the First 21 Days of Treatment
Description: Among the subjects treated with TMP (Paclitaxel/Margetuximab/Pertuzumab), report the number of subjects with dose-limiting toxicities (DLTs) during the first 21 days of treatment, where 21 days equals one cycle of treatment. DLTs are defined in Section 5.4 of the protocol, with the specified toxicities and lab values categorized and graded according to CTCAE v5.0.
Time Frame: From first treatment to 21 days
Population: All subjects treated at least one dose of TMP (Paclitaxel/Margetuximab/Pertuzumab).
Measure: Count of Participants; unit: Participants
Groups:
- Paclitaxel + Pertuzumab + Margetuximab: The research study procedures include screening for eligibility and study treatment including laboratory evaluations, two mandatory research biopsies and follow up visits. Cycle=21 days
  Paclitaxel- via IV, Day 1,8,15 of each cycle Margetuximab via IV, Day 1 of each cycle Pertuzumab via IV, Day 1 of each cycle
  Paclitaxel: Pre-determined dose administered via IV, Day 1,8,15 of each cycle 4 study cycles, or 12 weeks.
  Pertuzumab: Pre-determined dose administered via IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
  Margetuximab: Pre-determined dose administered by IV - Day 1 of each 21- day cycle 4 study cycles, or 12 weeks.
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab
Number analyzed (Participants) | 117
Participants
  Dose-limiting toxicity observed | 2
  Dose-limiting toxicity not observed | 115

8. Secondary Outcome: Maximum Grade of All Treatment-related Adverse Events During Neoadjuvant Treatment
Description: Maximum grade of all treatment-related adverse events (TRAEs) according to CTCAE v5.0 during neoadjuvant treatment, recorded per patient per arm. Subjects with no TRAEs reported (Grade 0) and Grade 1 adverse events are combined into a single category because only adverse events of Grade 2 or more were consistently reported.
Time Frame: Time from first dose of neoadjuvant treatment to start of de-escalated MP or HP protocol adjuvant therapy if subject received the de-escalated MP or HP protocol adjuvant therapy, up to 1 year after the last dose of their neoadjuvant treatment.
Population: All subjects who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
Number analyzed (Participants) | 117 | 54
Participants
  Grade 0 (no toxicities reported) or 1 (mild) | 23 | 16
  Grade 2 (moderate) | 68 | 24
  Grade 3 (severe) | 25 | 14
  Grade 4 (life threatening) | 1 | 0
  Grade 5 (fatal) | 0 | 0

9. Secondary Outcome: Patient-reported Outcomes
Description: Patient-reported outcomes for symptoms and quality of life (both physical and mental health) during neoadjuvant TMP and THP
Time Frame: From first treatment to 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Event-free Survival Rate (EFS)
Description: The distribution of the survival function and cumulative incidence function for EFS, summarized using the Kaplan Meier product limit estimator and 90% confidence interval (CI) using Greenwood's formula for the standard error
Time Frame: From enrollment to occurrence invasive local/regional recurrence distant recurrence or death from breast cancer or up to 10 years
Reporting Status: Not Posted

11. Secondary Outcome: Event-free Survival Rate (EFS) Patients With RCB 0 or 1
Description: as for outcome 10
Time Frame: From enrollment to occurrence of invasive local/regional recurrence distant recurrence or death from breast cancer or up to 10 years
Reporting Status: Not Posted

12. Secondary Outcome: Event-free Survival Rate (EFS)Patients With RCB 2 or 3
Description: as for outcome 10
Time Frame: as for outcome 11
Reporting Status: Not Posted

13. Secondary Outcome: Event-free Survival Rate (EFS) Patients Randomized to Neoadjuvant TMP
Description: as for outcome 10
Time Frame: as for outcome 11
Reporting Status: Not Posted

14. Secondary Outcome: Event-free Survival Rate (EFS) Patients Randomized to Neoadjuvant THP
Description: as for outcome 10
Time Frame: as for outcome 11
Reporting Status: Not Posted

15. Secondary Outcome: Event-free Survival Rate (EFS) -Patients With pCR
Description: as for outcome 10
Time Frame: as for outcome 11
Reporting Status: Not Posted

16. Secondary Outcome: Event-free Survival Rate (EFS) -Patients Without pCR
Description: as for outcome 10
Time Frame: as for outcome 11
Reporting Status: Not Posted

17. Secondary Outcome: Recurrence-free Interval Rate (RFI)
Description: The distribution of the survival function and cumulative incidence function for RFI summarized using the Kaplan Meier product limit estimator and 90% confidence interval (CI) using Greenwood's formula for the standard error
Time Frame: patients who undergo surgery for breast cancer as the interval from the time of surgery until the occurrence of invasive local/regional recurrence distant recurrence or death from breast cancer or up to 10 years
Reporting Status: Not Posted

18. Secondary Outcome: Recurrence-free Interval Rate (RFI) RCB 0 or 1
Description: as for outcome 17
Time Frame: as for outcome 17
Reporting Status: Not Posted

19. Secondary Outcome: Recurrence-free Interval Rate (RFI) RCB 2 or 3
Description: as for outcome 17
Time Frame: as for outcome 17
Reporting Status: Not Posted

20. Secondary Outcome: Recurrence-free Interval Rate (RFI) Patients Randomized to Neoadjuvant TMP
Description: as for outcome 17
Time Frame: as for outcome 17
Reporting Status: Not Posted

21. Secondary Outcome: Recurrence-free Interval Rate (RFI) Patients Randomized to Neoadjuvant THP
Description: as for outcome 17
Time Frame: as for outcome 17
Reporting Status: Not Posted

22. Secondary Outcome: Recurrence-free Interval Rate (RFI) Patients With pCR
Description: as for outcome 17
Time Frame: patients who undergo surgery for breast cancer as the interval from the time of surgery until the occurrence of invasive local/regional recurrence distant recurrence ror death from breast cancer or up to 10 years
Reporting Status: Not Posted

23. Secondary Outcome: Recurrence-free Interval Rate (RFI) Patients Without pCR
Description: as for outcome 17
Time Frame: as for outcome 17
Reporting Status: Not Posted

24. Secondary Outcome: Overall Survival Rate (OS)
Description: The distribution of the survival function and cumulative incidence function for OS, summarized using the Kaplan Meier product limit estimator and 90% confidence interval (CI) using Greenwood's formula for the standard error
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

25. Secondary Outcome: Overall Survival Rate (OS) Patients With RCB 0 or 1
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

26. Secondary Outcome: Overall Survival Rate (OS) Patients With RCB 2 or 3
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

27. Secondary Outcome: Overall Survival Rate (OS) Patients Randomized to Neoadjuvant TMP
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

28. Secondary Outcome: Overall Survival Rate (OS) Randomized to Neoadjuvant THP
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

29. Secondary Outcome: Overall Survival Rate (OS) Patients With pCR
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

30. Secondary Outcome: Overall Survival Rate (OS) Patients Without CR
Description: as for outcome 24
Time Frame: up to 10 years from definitive surgery.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time from first dose of neoadjuvant treatment to start of de-escalated MP or HP protocol adjuvant therapy if subject received the de-escalated MP or HP protocol adjuvant therapy, up to 1 year after the last dose of their neoadjuvant treatment.
Description: Regular investigator assessment
Arm/Group | Paclitaxel + Pertuzumab + Margetuximab | Paclitaxel + Pertuzumab + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 1/117 | 0/54
Serious Adverse Events (participants affected / at risk) | 4/117 | 1/54
Other Adverse Events (participants affected / at risk) | 105/117 | 46/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Pertuzumab + Margetuximab (N=117) | Paclitaxel + Pertuzumab + Trastuzumab (N=54)
Catheter related infection (Infections and infestations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Pertuzumab + Margetuximab (N=117) | Paclitaxel + Pertuzumab + Trastuzumab (N=54)
Anemia (Blood and lymphatic system disorders) | 22 | 16
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Blurred vision (Eye disorders) | 3 | 3
Dry eye (Eye disorders) | 6 | 1
Flashing lights (Eye disorders) | 1 | 1
Floaters (Eye disorders) | 1 | 1
Vision decreased (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Belching (Gastrointestinal disorders) | 1 | 1
Bloating (Gastrointestinal disorders) | 8 | 1
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhea (Gastrointestinal disorders) | 48 | 23
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 9 | 4
Dysphagia (Gastrointestinal disorders) | 12 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 9 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 23 | 3
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 6 | 13
Oral pain (Gastrointestinal disorders) | 6 | 1
Periodontal disease (Gastrointestinal disorders) | 6 | 1
Stomach pain (Gastrointestinal disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5
Edema limbs (General disorders) | 2 | 2
Fatigue (General disorders) | 31 | 10
Fever (General disorders) | 2 | 1
Flu like symptoms (General disorders) | 1 | 1
Generalized edema (General disorders) | 1 | 1
Localized edema (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 5 | 3
Pain (General disorders) | 5 | 1
Allergic reaction (Immune system disorders) | 0 | 2
Anaphylaxis (Immune system disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 2 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2
Otitis externa (Infections and infestations) | 3 | 1
Papulopustular rash (Infections and infestations) | 8 | 2
Rash pustular (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 1
Thrush (Infections and infestations) | 1 | 2
Upper respiratory infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 4
Vaginal infection (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 6 | 1
Thrush (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 5 | 1
Vaginal infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 9
Seroma (Injury, poisoning and procedural complications) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 32 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 13 | 9
Alkaline phosphatase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 8 | 8
Blood bilirubin increased (Investigations) | 3 | 1
CD4 lymphocytes decreased (Investigations) | 3 | 1
Creatinine increased (Investigations) | 10 | 1
Ejection fraction decreased (Investigations) | 18 | 1
Lymphocyte count decreased (Investigations) | 1 | 6
Lymphocyte count increased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 8 | 10
Weight gain (Investigations) | 8 | 1
Weight loss (Investigations) | 8 | 3
White blood cell decreased (Investigations) | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 7
Hypernatremia (Metabolism and nutrition disorders) | 6 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 7 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 5 | 6
Headache (Nervous system disorders) | 8 | 6
Memory impairment (Nervous system disorders) | 12 | 1
Paresthesia (Nervous system disorders) | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 11
Paresthesia (Nervous system disorders) | 6 | 11
Peripheral motor neuropathy (Nervous system disorders) | 2 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 11
Tremor (Nervous system disorders) | 1 | 11
Anxiety (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 7 | 3
Irritability (Psychiatric disorders) | 1 | 3
Dysuria (Renal and urinary disorders) | 1 | 3
Glucosuria (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 1
Amenorrhea (Reproductive system and breast disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 7 | 3
Irregular menstruation (Reproductive system and breast disorders) | 1 | 1
Vaginal dryness (Reproductive system and breast disorders) | 1 | 1
Vaginal pain (Reproductive system and breast disorders) | 1 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 1
Vaginal pain (Reproductive system and breast disorders) | 2 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 11
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 5
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 9
Scalp pain (Skin and subcutaneous tissue disorders) | 2 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 20 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 11 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 2 | 3
Hot flashes (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 11 | 16
Thromboembolic event (Vascular disorders) | 12 | 1
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04425018/Prot_SAP_000.pdf